CLINICAL TRIAL: NCT06792500
Title: Investigational Study of Glycerol Tributyrate in MELAS and LHON-Plus
Brief Title: A Basket Clinical Study to Assess Glycerol Tributyrate in Patients With Mitochondrial Encephalopathy, Lactic Acidosis, Stroke-like Episodes (MELAS) or Leber's Hereditary Optic Neuropathy-Plus (LHON-Plus)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001021; UH3TR003897 (NIH)
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: MELAS Syndrome; Lebers Hereditory Optic Neuropathy With Extra Ocular Symptoms (LHON-Plus)
Keywords: Mitochondrial Disease; Pathogenic mitochondrial variants; ATP deficiency; Maternal inheritance; Stroke-like episodes; Chronic energy deficit; Deficient oxidative phosphorylation; Seizures; Extreme tiredness; Myopathy; Migraines; Gastrointestinal dysmotility; visual loss; Dystonia; Anxiety; Hearing loss; Tremors; Lactic Acidosis; Cognitive deficit; Neuropathy; m.3243 variant; m.11778 variant
MeSH Terms: conditions — MELAS Syndrome; Mitochondrial Diseases; Seizures; Muscular Diseases; Migraine Disorders; Vision Disorders; Dystonia; Anxiety Disorders; Hearing Loss; Tremor; Acidosis, Lactic; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MELAS (Experimental): 12 MELAS participants will be enrolled in the baseline phase before being given an oral administration of glycerol tributyrate. All participants will undergo a six-month-long non-randomized dose escalation phase to determine each participant-specific maximum tolerated dose (MTD), after which the fixed MTD of glycerol tributyrate will be orally administered during the 12-month-long clinical phase.
  Interventions: Drug: Glycerol Tributyrate
- LHON-Plus (Experimental): 12 LHON-Plus participants will be enrolled and will be given the interventional drug, glycerol tributyrate. All participants will undergo a six-month-long non-randomized dos escalation phase in order to determine the patient-specific maximum tolerated dose (MTD), after which they will be orally administered this MTD for a period of 12 months.
  Interventions: Drug: Glycerol Tributyrate

INTERVENTIONS:
Drug: Glycerol Tributyrate — Participants will be administered orally three times a day enteric hard capsules containing 500 mg of glycerol tributyrate with an 8-ounce glass of water on an empty stomach: morning, noon, and evening during the dose-escalation phase. Each MELAS participant will undergo a six-month dose escalation phase of glycerol tributyrate, starting at a dose of 1,000 mg (tid) per day during the first month followed by a monthly increase of 500 mg (tid) per dose of glycerol tributyrate with the maximal oral dose of glycerol tributyrate 3,500 mg (tid) per dose at the end of six-month-long dose escalation phase. Once the participant-specific fixed maximum tolerated dose (MTD) is determined, MELAS participants will take an oral administration of this MTD three times a day during the 12-month-long clinical phase.

SUMMARY:
This is a parallel arm non-randomized dose-escalation, open-label basket exploratory phase 1 clinical trial where Mitochondrial encephalopathy, lactic acidosis, stroke-like episodes (MELAS) and Leber's hereditary optic neuropathy-Plus (LHON-Plus) participants will undergo simultaneous enrollment in two disease-based arms and receive daily oral doses of glycerol tributyrate to assess its safety and potential for efficacy using clinical, biochemical, and molecular evidence.

This study will utilize a two-month baseline lead-in phase to establish and document the clinical baseline for each participant in both arms in order to compare the molecular and clinical parameters. This is clinically relevant in light of the high clinical heterogeneity among subjects affected by the same mitochondrial disease (MELAS or LHON-Plus). For ethical concerns prompted by the lack of treatment for these two intractable and progressive mitochondrial diseases, there will not be a placebo control group. Thus, each participant will act as their own control and receive oral doses of glycerol tributyrate, eliminating the need for a placebo. Considering the high clinical heterogeneity among participants affected by MELAS or LHON-Plus and some clinical divergence between MELAS and LHON-Plus, this strategy is beneficial to every enrolled participants, as each will receive the investigational drug, glycerol tributyrate. In addition, this approach will determine the subject-specific maximal optimized dose in a personalized medicine-based approach.

After approval of the IRB protocol from the Institutional Review Board Data and signed consent form from all participants, this investigational basket clinical trial has three phases spanning over 20 months:

* A baseline lead-in phase (2 months) to collect participant-specific baseline for clinical, biochemical, molecular and metabolic biomarkers that will be monitored throughout the subsequent dose-escalation and clinical phases.
* A dose-escalation phase (6 months) to determine the participant-specific maximum tolerated dose (MTD) during which participant-specific clinical and biochemical biomarkers are collected every month.
* A clinical phase at a fixed subject-specific MTD dose (12 months) to collect participant-specific clinical, biochemical, molecular and metabolic biomarkers and to perform three scheduled skin biopsies: at the outset, mid-point, and the end of this clinucal phase. We have planned for a 12-month-long clinical phase at a fixed participant-specific MTD considering the absence of reliable predictors that makes idiosyncratic disease-specific symptoms for MELAS and LHON-Plus impossible to forecast among participant for assessing the potential efficacy of glycerol tributyrate by monitoring clinical symptoms specific for each disease. During the 12-month-long time-frame, disease-specific clinical symptoms will be collected as preliminary evidence of efficacy of glycerol tributyrate using disease-specific biomarkers.

Finally, discharge procedure during which the clinical investigator will record non-serious adverse events or serious adverse events for 7 or 30 days, respectively, after the last day of study participation.

DETAILED DESCRIPTION:
During the two-month-long baseline lead-in phase, we will acquire the following information, which are part of standard clinical care:

1. Medical history
2. Pregnancy test for subjects of childbearing potential: using a urine human chorionic gonadotropin test
3. Number of hospitalizations in the last 12 months
4. Physical examination
5. 6-minute-walk test
6. Clinical laboratory biomarkers completed and/or interpreted at the CLIA-certified labs at Children's National Hospital:

   * GDF-15
   * FGF-21
   * CMP
   * Hemoglobin A1C
   * Plasma amino acids
   * Lactate
   * Carnitine and acylcarnitine
   * Urine organic acids and urine analysis
7. Standard 1 hour-long EEG for MELAS subjects
8. Baseline MRI (for subjects with MELAS or LHON-Plus) and MRS (for MELAS subjects)
9. Screen for stroke-like episodes for MELAS subjects
10. Electronic seizure diary for MELAS subjects
11. Motor examination for subjects with MELAS or LHON-Plus
12. Electromyography and nerve conduction velocity for LHON-Plus subjects
13. Ophthalmological examination (fundi, visual field, and visual acuity) for LHON-Plus subjects
14. Snellen chart exam for LHON-Plus subjects
15. Lumbar puncture for LHON-Plus subjects to assess CSF markers for multiple sclerosis-like:

    * A specific group of antibodies referred to as oligoclonal bands
    * Myelin basic proteins (MBP)
    * IgG levels
    * Levels of inflammasome proteins
    * Leukocytes count: lymphocytes (B-cells and T-cells), monocytes, macrophages, plasma cells, and granulocytes
    * CSF/serum glucose ratio
16. Fatigue screen using the Modified Fatigue Impact Scale
17. Quality of Life (QoL) is assessed using the short questionnaire "Neuro-Quality of life"
18. Cognitive assessment using the NIH-Toolbox Cognitive Battery
19. Skin biopsy to assess:

    * Mitochondrial Genetic Analysis: Quantification of the heteroplasmic levels of MELAS and LHON-Plus mitochondrial variants by long-range PCR followed by massively parallel sequencing done at Baylor Miraca Genetics Laboratories DBA Baylor Genetics, Clinical Diagnostics Laboratory.
    * Mitochondrial Respiratory Chain Enzyme Analysis: Quantification of enzymatic activity of oxidative phosphorylation (OXPHOS) Complexes by spectrophotometry done by Baylor Genetics.
    * Mitochondrial Fitness Assays: The mitochondrial fitness of participant-derived dermal fibroblasts are assessed in real-time by live-cell mitochondrial assays using the two world's most advanced automated cell metabolism analyzers and the automated normalization system, Cytation1, from Agilent Technologies Inc., and the three following specialized metabolic assays from Agilent:

Mitochondrial Stress Test assay: This assay measures the baseline of the participant's mitochondrial functions by quantifying OXPHOS bioenergetic parameters. The investigators uses this assay to monitor the potential efficacy of oral administration of glycerol tributyrate in participants.

Real-Time ATP Rate assay: The investigators use this assay to quantify the pathway-specific ATP rate production from the mitochondrial OXPHOS pathway and the cytosolic glycolytic pathway.

Agilent Glycolytic Rate assay: The investigators use this assay to assess the metabolic plasticity between the two main energy pathways, OXPHOS and glycolysis,as well as to correlate one-on-one the glycolytic activity with lactate accumulation.

No participants are enrolled in the dose-escalation phase without a complete interpretation of the clinical data from the baseline lead-in phase. As a higher level of safety risk, participants with the pre-existing severe complications, renal failure, arrhythmia, pneumonia with respiratory failure, and/or severe gastroparesis, will be excluded from progressing to the dose-escalating phase.

During the six-month-long dose-escalation phase, the investigators will determine the safe participant-specific MTD using the toxicology and clinical data described above.

Participants are administered glycerol tributyrate three times a day (tid) dispensed by the Children's National Hospital (CNH) research pharmacy located in the study site (CNH). To initiate the dose-escalation phase, the investigator provides all participants with a one-month supply of 100 capsules, each containing 500 mg of glycerol tributyrate. The initial dose is 1000 mg tid. During the last week of month 1 and subsequent months, the investigators review the clinical and biochemical data for each participant before increasing the oral dose of glycerol tributyrate.

Below is the description of the methods to assess for dose-limiting toxicity (DLT) throughout the dose-escalation phase.

1. Disease-specific assessment:

   * For participants with MELAS, there are two measurable and reliable biomarkers for MELAS-specific upper threshold of the effect of the investigational drug: 1) plasma lactate levels greater than three times the normal levels; and 2) blood glucose levels above 200 mg/dl (11.1 mM). In addition, general toxicity is assessed in participants with MELAS as described in the criteria detailed below, which are shared by all participants. If general toxicity and/or MELAS-specific upper threshold of plasma lactate levels and blood glucose levels, MELAS participants will not be escalated to the next planned dose by 500 mg tid but rather re-treated at a one-dose concentration lower than the dose at which Grade 3 toxicity is encountered.
   * For participants with LHON-Plus, there are no similar reliable biomarkers for assessing such upper threshold. Therefore, these subjects will be closely monitored for general toxicity.
2. General toxicity assessment: The clinical investigators evaluate toxicity using the Common Terminology Criteria of Adverse Events (CTCAE) version 4.0 3 grading scale.

   * Dose-limiting toxicity (DLT) is defined as any of the adverse effects (AE) listed in Section 5.3.1.11 "Toxicity Monitoring" graded on the CTCAE v4.03. AE is considered possibly related to the investigational drug that occurs any time from the initial dose of glycerol tributyrate, when at grade 3 or higher, or worsening of baseline status as defined by increase of at least 2 grades, if baseline grade is less than or equal to 1. participants who develop Grade 3 or higher toxicity are re-treated at a one-dose concentration lower than the dose at which Grade 3 toxicity is encountered.
   * In the absence of DLT or in the case of CTCAE grade 1 or 2 toxicity, dose of glycerol tributyrate is escalated to the next planned dose by 500 mg tid. Doses are increased to the next planned dose by 500 mg tid every month until month 6 or prior if the participant-specific DLT is reached based on toxicity data using the CTCAE grading scale, as defined above. If participants reach their MTD prior to month 6 of the dose-escalating phase, they immediately enter the clinical phase at the fixed participant-specific MTD, defined as a one-dose concentration lower than the dose at which Grade 3 toxicity is encountered.

At the conclusion of the dose-escalation phase, a skin biopsy will be performed on all participants prior to the onset of the clinical phase at fixed participant-specific MTD. The participant-specific dermal fibroblasts will be derived to determine the genetic and mitochondrial bioenergetic parameters for each participant at the outset of the clinical phase.

The 12 month-long clinical phase at fixed participant-specific MTD starts at the conclusion of the 6-month-long dose-escalation phase and is divided into two 6-month-long periods. This 12-month-long time-frame is necessary to capture disease-specific clinical symptoms, to collect preliminary evidence of efficacy of glycerol tributyrate using disease-specific biomarkers, and to assess possible clinical outcomes demonstrating clinical benefit of glycerol tributyrate.

At the outset, mid-phase, and end of the 12 month-long clinical phase, participants will undergo three skin biopsies to assess the potential efficacy of glycerol tributyrate on:

1. OXPHOS bioenergetic parameters
2. the clinical and biochemical target biomarkers.

Throughout the clinical phase at fixed MTD, we will implement the same safety assessment for DLTs than for the dose-escalation phase.

At the end of the 12-month-long clinical phase at fixed participant-specific MTD, the investigators will discharge the participants after performing a follow-up study during which non-serious adverse events or serious adverse events will be recorded for 7 or 30 days, respectively, after the last day of study participation.

Capsules containing glycerol tributyrate (500 mg) will be administered orally to all participants three times a day with an 8-ounce glass of water on an empty stomach: morning, noon, and evening during the dose-escalation phase and the clinical phase at fixed subject-specific MTD of the study.

Compliance will be assessed with an electronic log/diary where participants will record on a daily basis time, date, and pill counts. Participants will be asked to bring back all the bottles of glycerol tributyrate to subsequent visits to assess compliance. Compliance will be considered satisfactory with 80% of planned doses logged in.

Participants will be specifically monitored for the occurrence of the following Adverse Events (AEs) graded based on the CTCAE v4.03:

* Dizziness
* Syncope
* Concentration impairment
* Fatigue
* Fever
* Nausea
* Vomiting
* Diarrhea
* Hypoglycemia
* Hyperglycemia
* Lactic acidosis The investigators will review any AEs in person during the scheduled visits. The participants will also fill out a survey on their electronic diary to make it easier to capture any AEs.

A Data and Safety Monitoring Board (DSMB) committee has been formed and includes five independent members: a metabolic physician, neurologist, bioethicist, a clinical trialist, and a lay person as a non-voting member. The DSMB committee will review safety data on an ongoing basis, meet biannually or ad-hoc if the need arises. This additional oversight provided by a DSMB committee provides further protection to the study participants during the basket clinical trial for MELAS and LHON-PLus.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 18 to 65 years
* A confirmed molecular diagnosis of MELAS or LHON-Plus
* Symptomatic participants with MELAS harboring the m.3243A>G variant or a mitochondrial pathogenic variant solely mapping in a mitochondrial gene encoding a mitochondrial subunit of Complex I
* Symptomatic participants with LHON-Plus harboring the m.11778G>A or a mitochondrial pathogenic variant only mapping in a mitochondrial gene encoding a mitochondrial subunit of Complex I
* Normal enzymatic Complex II activity
* Participants able to swallow capsules and comply with the requirements of the study according to the opinion of the investigator
* Able to give written, informed consent
* Participants who are sexually active and/or fertile must use an effective birth control during the study

Exclusion Criteria:

* • History of another primary mitochondrial disorder

  * Participants acutely ill
  * Positive urine pregnancy test for female subjects of childbearing potential within seven days prior to the first dose of the investigational drug
  * Pregnancy and/or breastfeeding
  * Participating in another mitochondrial disorder trial
  * Participated in another mitochondrial disorder trial within the last six months
  * On a current therapy with other investigational agents
  * Absence of neurological symptoms, muscle weakness, or exercise intolerance
  * Presence of any of the following signs or symptoms in the past six months at grade 3 or higher based on the CTCAE version 4.03: nausea, vomiting, diarrhea, hypoglycemia, hyperglycemia, dizziness, blurred vision, or syncope
  * A known hypersensitivity to any excipient contained in the drug formulation
  * Current abuse of drugs and/or alcohol
  * Unable to consent for themselves
  * Participants with an enteral feeding tube
  * Inability to travel to the study site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of Dose Safety for Glycerol Tributyrate | 20 months
  To assess the dose safety of the investigational drug, glycerol tributyrate, the investigators will measure Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] using the CTCAE version 4.03
Potential Efficacy of Glycerol Tributyrate on the oxidative phsophorylation metabolism | 20 months
  The investigators will assess whether participant-specific maximum tolerated dose (MTD) of glycerol tributyate results in increase of the participant's bioenergetic parameters for the oxidative phosphorylation pathway and/or mitochondrial ATP rate production above the participant's baseline determined from a dermal fibroblasts derive from a skin biopsy during the two-month-long baseline lead-in phase.

SECONDARY OUTCOMES:
Shared Secondary MELAS and LHON-Plus Outcome | 20 months
  Improved daily activity measured by actigraphy
Shared Secondary MELAS and LHON-Plus Outcome | 20 months
  Improved performance in the 6-minute-walking test
Shared Secondary MELAS and LHON-Plus Outcome | 20 months
  Reduced frequency of hospitalization prior to trial entry
Shared Secondary MELAS and LHON-Plus Outcome | 20 months
  Improved quality of life (QoL) using the Neuro-QoL
Shared Secondary MELAS and LHON-Plus Outcome | 20 months
  Reduced presence and perceived fatigue using the Modified Fatigue Impact Scale
MELAS-Specific Secondary Outcome Measure | 20 months
  Decreased frequency of seizures
MELAS-Specific Secondary Outcome Measure | 20 months
  Stable cortical brain lesions by magnetic resonance imaging
LHON-Plus Specific Secondary Outcome Measure | 20 months
  Stable hemoglobin A1C
LHON-Plus Specific Secondary Outcome Measure | 20 months
  Stable brain and spinal lesions by magnetic resonance imaging
LHON-Plus Specific Secondary Outcome Measure | 20 months
  Stable cerebrospinal fluid markers for Multiple Sclerosis-like presentations

OTHER OUTCOMES:
MELAS-Specific Exploratory Outcome | 20 months
  Decreased blood and brain lactate levels, measured by plasma and magnetic resonance spectroscopy, respectively.
MELAS-Specific Exploratory Outcome | 20 months
  Stable cortical brain lesions by magnetic resonance imaging
LHON-Plus-Specific Exploratory Outcome | 20 months
  Improved visual acuity measured by Snellen chart
LHON-Plus Specific Exploratory Outcome Measure | 20 months
  Improved electromyography and nerve conduction velocity
LHON-Plus-Specific Exploratory Outcome Measure | 20 months
  Decreased Multiple Sclerosis-like presentations using the Expanded Disability Status Scale

CONTACTS AND LOCATIONS:
Overall Officials: Debra Regier, M.D., Ph.D., Principal Investigator — Children's National Hospital; Children's National Rare Disease Institute; Wei-Liang Chen, M.D., Study Chair — Children's National Research Institute; Anne Chiaramello, Ph.D., Study Director — George Washington University School of Medicine and Health Sciences
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No